CLINICAL TRIAL: NCT03297541
Title: Healthy Kids at I-PAL (Interactive Physical Activity Lab)
Brief Title: Healthy Kids I-PAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Southeastern Louisiana University (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2016-009
Record Dates: First submitted 2017-09-18; First posted 2017-09-29 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- m-health approach (Experimental): All dyads will receive the m-health approach.
  Interventions: Behavioral: m-health approach

INTERVENTIONS:
Behavioral: m-health approach — Parent/child dyads attend remote counseling sessions delivered over Internet-connected device (e.g. smartphone, iPad/tablet, laptop, or desktop computer). A counselor will deliver the lesson, review progress based on the objectively measured data, and provide individualized advice and problem-solving strategies for parent and child. Families will receive weekly contact via smartphone. Each lesson will include an interactive component for parent and child related to healthy eating and active play, as well as an interactive parenting training component. Lessons are based on the family treatment methods that effectively promote child and parent weight loss that is sustained for 10 years (Epstein et al., 1990; Epstein et al., 1981). Anthropometric and demographic data collected on children in the dyad only.

SUMMARY:
Up to 30 parent/child dyads will be recruited to participate in an m-Health intervention (delivered over smartphone, iPad/Tablet, or desktop/laptop) to promote healthy behaviors and healthy weight among children and their parents.

ELIGIBILITY:
Inclusion Criteria for Child:

* Have at least one participating parent
* Be physically capable of exercise
* Be free of diseases that affect metabolism, body weight, and food intake, including type 1 or type 2 diabetes, HIV/AIDS, and cancer

Inclusion Criteria for Parent:

* Have a smart phone
* Be willing to use the smartphone for the mHealth intervention

Exclusion Criteria for Child:

* Significant cardiovascular disease or disorders via self-report from parent
* Other significant medical problems that would prevent them from engaging in regular physical activity.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Staiano, PhD, Principal Investigator — Pennington Biomedical Research Center; Corby Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Southeastern Louisiana University, Hammond, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staiano AE, Shanley JR, Kihm H, Hawkins KR, Self-Brown S, Hochsmann C, Osborne MC, LeBlanc MM, Apolzan JW, Martin CK. Digital Tools to Support Family-Based Weight Management for Children: Mixed Methods Pilot and Feasibility Study. JMIR Pediatr Parent. 2021 Jan 7;4(1):e24714. doi: 10.2196/24714. PMID 33410760

RESULTS

PARTICIPANT FLOW:
Groups:
- M-health Approach: All dyads will receive the m-health approach.
  m-health approach: Parent/child dyads attend remote counseling sessions delivered over Internet-connected device (e.g. smartphone, iPad/tablet, laptop, or desktop computer). A counselor will deliver the lesson, review progress based on the objectively measured data, and provide individualized advice and problem-solving strategies for parent and child. Families will receive weekly contact via smartphone. Each lesson will include an interactive component for parent and child related to healthy eating and active play, as well as an interactive parenting training component. Lessons are based on the family treatment methods that effectively promote child and parent weight loss that is sustained for 10 years (Epstein et al., 1990; Epstein et al., 1981).
Period: Overall Study
Arm/Group | M-health Approach
Started | 10 (10 children and 10 parents)
Completed | 10 (10 children and 10 parents)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics data were collected from the children in the dyads only.
Groups:
- Child Participants in the Dyads: All dyads will receive the m-health approach.
  m-health approach: Parent/child dyads attend remote counseling sessions delivered over Internet-connected device (e.g. smartphone, iPad/tablet, laptop, or desktop computer). A counselor will deliver the lesson, review progress based on the objectively measured data, and provide individualized advice and problem-solving strategies for parent and child. Families will receive weekly contact via smartphone. Each lesson will include an interactive component for parent and child related to healthy eating and active play, as well as an interactive parenting training component. Lessons are based on the family treatment methods that effectively promote child and parent weight loss that is sustained for 10 years (Epstein et al., 1990; Epstein et al., 1981).
Arm/Group | Child Participants in the Dyads
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Child Acceptability of the mHealth Approach
Description: Children completed an acceptability survey at the end of the intervention that included Likert scales on intervention satisfaction. The items were average to calculate an average acceptability score. The scale range for the average total score is 1 to 5. A higher score indicates higher acceptability.
Time Frame: 13 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | M-health Approach
Number analyzed (Participants) | 10
score on a scale | 3.8 (.5)

2. Secondary Outcome: BMI Z-score Change
Description: Objectively measured height and weight were compared against the normative values for age (months) and sex according to the CDC growth charts. A z-score is assigned, with 0 representing the population mean. A positive z-score indicates a BMI above the population mean (higher relative weight), whereas a negative z-score is below the population mean (lower relative weight). For the change score, the post BMI z-score measured at week 14-16 was subtracted from the baseline BMI z-score. For the change score, a positive value indicates an increase in relative weight, whereas a negative value indicates a reduction in relative weight.
Time Frame: Week 0 to Week 14-16
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- Child: All dyads will receive the m-health approach.
  m-health approach: Parent/child dyads attend remote counseling sessions delivered over Internet-connected device (e.g. smartphone, iPad/tablet, laptop, or desktop computer). A counselor will deliver the lesson, review progress based on the objectively measured data, and provide individualized advice and problem-solving strategies for parent and child. Families will receive weekly contact via smartphone. Each lesson will include an interactive component for parent and child related to healthy eating and active play, as well as an interactive parenting training component. Lessons are based on the family treatment methods that effectively promote child and parent weight loss that is sustained for 10 years (Epstein et al., 1990; Epstein et al., 1981).
Arm/Group | Child
Number analyzed (Participants) | 10
Z-Score | -0.14 (0.17)

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: Children & Parents in dyads;
Groups:
- Parent Participants in the Dyads: All dyads will receive the m-health approach.
  m-health approach: Parent/child dyads attend remote counseling sessions delivered over Internet-connected device (e.g. smartphone, iPad/tablet, laptop, or desktop computer). A counselor will deliver the lesson, review progress based on the objectively measured data, and provide individualized advice and problem-solving strategies for parent and child. Families will receive weekly contact via smartphone. Each lesson will include an interactive component for parent and child related to healthy eating and active play, as well as an interactive parenting training component. Lessons are based on the family treatment methods that effectively promote child and parent weight loss that is sustained for 10 years (Epstein et al., 1990; Epstein et al., 1981).
Arm/Group | Child Participants in the Dyads | Parent Participants in the Dyads
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
A limitation of these studies is the one-arm design without a control or comparator and the need for further verification in a larger randomized controlled trial. It is possible that BMIz fluctuations were influenced by maturation bias or regression to the mean, though the observed effect size was similar to prior interventions. Another limitation is the use of BMIz to examine change, as researchers have identified concerns with z-score for children with a BMI above the 97th percentile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03297541/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03297541/SAP_001.pdf
  • Informed Consent Form (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03297541/ICF_002.pdf